CLINICAL TRIAL: NCT00305968
Title: Evaluation of Patient Education in Patients With Irritable Bowel Syndrome - a Randomized Multi Center Study
Brief Title: Evaluation of Patient Education in Irritable Bowel Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: Sykehuset Telemark (Other Government); The Hospital of Vestfold (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SSHFIBS-1
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Irritable Bowel Syndrome
Keywords: Quality of life; Gastrointestinal symptoms; Health related costs
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Patient Education as Topic

INTERVENTIONS:
Behavioral: patient education — Patient education group

SUMMARY:
About 10% of the population in western countries suffer from abdominal pain and change of bowel habits - known as the irritable bowel syndrome. The patients suffer from low quality of life and they are often not well taken care of within the public healthcare system. They often feel frustrated and seek both their family doctors, specialists and alternative medicine for help. Many patients feel they do not know enough about their disease, and the uncertainty may enhance bowel symptoms. We want to evaluate the effect of patient information and education in these patients.

DETAILED DESCRIPTION:
The patients are enrolled in endoscopic clinics in 7 hospitals in Norway. They are randomized to receive intervention now (intervention group) or in 6 months (control group). The intervention is a 6 hour education about the irritable bowel syndrome, held by a experienced gastroenterologist at the local hospital.

Elements in this "school-day" includes symptoms, epidemiology, pathophysiology, treatment, nutritional advices.

The patients are evaluated at time: 0 months and 6 months (intervention group and control group), 12 months (control group) and after 2 years (both groups).

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Irritable Bowel Syndrome, verified by the Rome II criteria
* Must be able to participate in a education-group

Exclusion Criteria:

* Another GI-diagnosis or kind of surgery that may interfere with the symptoms of irritable bowel syndrome
* Serious, untreated psychiatric disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Change in Quality of life | 6 months
Change in Gastrointestinal symptom score | 6 months

SECONDARY OUTCOMES:
Change in health related costs | 6 months
Evaluation of further patient needs after education | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jostein Sauar, PhD, Study Director
Locations (1):
- Sorlandet Sykehus HF, Kristiansand, Norway